CLINICAL TRIAL: NCT04580030
Title: Tricuapid Annular Plane Sistolic Excursion Before General Anesthesia Can Predict Hypotension After Induction
Acronym: (Tapse)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Bursa City Hospital (Other Government)
Responsible Party: Principal Investigator, Ferdi GÜLAŞTI, M.D. Specialist of anesthesiology and reanimation, Bursa City Hospital
Other Study IDs: 2020-6/1
Record Dates: First submitted 2020-10-02; First posted 2020-10-08 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Anesthesia
Keywords: General anesthesia; tricuspid anular plane systolic excursion; hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hypotension: Basal hemodynamic parameters and hemodynamic values will be taken every two minutes after induction until surgical incision. Patients with systolic pressure <90 mmHg or 30% drop in baseline, and mean artery pressure below 60 mmHg will be considered to have hypotension. Patients will be divided into two groups as "Hypotension" and "No Hypotension".
- no hypotension: Basal hemodynamic parameters and hemodynamic values will be taken every two minutes after induction until surgical incision. Patients with systolic pressure <90 mmHg or 30% drop in baseline, and mean artery pressure below 60 mmHg will be considered to have hypotension. Patients will be divided into two groups as "Hypotension" and "No Hypotension".

SUMMARY:
the investigators purpose is to predict hypotensive condition that can develop after general anesthesia induction by measuring the Tricuspid Annular Plane Systolic Movement (TAPSE), which is an echocardiographic parameter.

DETAILED DESCRIPTION:
Intraoperative hypotension development might increase myocardial damage, acute kidney damage, and septic complications, and have an effect on mortality increase. For this reason, prevention of an unwanted hypotensive event has an important role in reducing mortality and morbidity. The prediction of the risk of hypotension is generally based on the evaluation of the comorbid status and volume status of patients .It is already known that right ventricular systolic dysfunction has prognostic value in various pathological cases. It is quite difficult to evaluate the RV function with echocardiography because of the complex geometry of RV. Although RV function has been evaluated only visually for many years, guidelines have been published as a result of recent studies by the American Society of Echocardiography. In this respect, abnormal RV function should be suspected when one of the criteria of S '<10 cm /s, TAPSE <16 mm, RVFAC <35%, or R-MPI (Tissue Doppler)> 0.55. Normal and abnormal function is distinguished more reliably when combining more than one RV function measures. TAPSE is a parameter with which the apex-basal shortening can be easily measured, providing specific data on global RV function. It depends less on optimal image quality than other RV function measurements, and is an easy-to-measure criterion. Low TAPSE is not very common; however, it was measured in people with no heart disease due to diagnostic misclassification and excessive ends of the normal spectrum. the investigators think that despite the lack of cardiac disease, cardiac reserve functions of each patient may have limits in terms of development of hypotension in general anesthesia induction. The investigators considered that TAPSE, which decreased within normal limits in patients without cardiac disease, could predict hypotension development in general anesthesia induction, and planned study for this purpose.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective surgery
* Patients who will receive general anesthesia
* Patients between 18-65 years of age
* Physical status I or II according to the American Society of Anesthetists (ASA) in preoperative evaluation
* Those without known heart disease
* Patients with TAPSE value above 1.6 cm

Exclusion Criteria:

* Patients under the age of 8 and over 65,
* Pregnant patients,
* Patients who refuse to participate in the study,
* ASA III and above,
* Patients with known heart disease,
* Patients with TAPSE value of less than 1.6 measured with Transthoracic Echocardiography will not be allowed to be included in the study.
* Patients with difficult airway management or difficult intubation will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It was planned that a total of 40 patients undergoing elective general surgery under general anesthesia with standard general anesthesia induction would be included in this prospective and observational study.
Sampling Method: Probability Sample
Enrollment: 7 (Estimated)
Dates: Start 2020-09-09 (Actual); Primary Completion 2021-09-09 (Estimated); Study Completion 2021-09-10 (Estimated)

PRIMARY OUTCOMES:
tricuspid anular plane systolic excursion(TAPSE) | TAPSE will be measured with Transthoracic Echocardiography about 30 minutes before the induction in the preoperative period.
  The investigators purpose is to predict hypotensive condition that can develop after general anesthesia induction by measuring the Tricuspid Annular Plane Systolic Movement (TAPSE), which is an echocardiographic parameter.

CONTACTS AND LOCATIONS:
Overall Officials: Ferdi Gülaştı, Study Chair — Bursa City Hospital
Locations (1):
- Bursa City Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Zhang J, Critchley LA. Inferior Vena Cava Ultrasonography before General Anesthesia Can Predict Hypotension after Induction. Anesthesiology. 2016 Mar;124(3):580-9. doi: 10.1097/ALN.0000000000001002. PMID 26771910
- [Result] Szabo M, Bozo A, Darvas K, Horvath A, Ivanyi ZD. Role of inferior vena cava collapsibility index in the prediction of hypotension associated with general anesthesia: an observational study. BMC Anesthesiol. 2019 Aug 7;19(1):139. doi: 10.1186/s12871-019-0809-4. PMID 31390983
- [Result] Main AB, Braham R, Campbell D, Inglis AJ, McLean A, Orde S. Subcostal TAPSE: a retrospective analysis of a novel right ventricle function assessment method from the subcostal position in patients with sepsis. Ultrasound J. 2019 Aug 27;11(1):19. doi: 10.1186/s13089-019-0134-7. PMID 31456096